CLINICAL TRIAL: NCT00256945
Title: In Vivo Study of the Relationship Between Surface Roughness of a Dental Restorative Material and Biofilm Formation
Brief Title: Surface Roughness of a Dental Restorative Material and Biofilm Formation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 191057HMO-CTIL
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2007-12

CONDITIONS: Diabetic; Antibiotic Intake
Keywords: biofilm formation; dental plaque; surface roughness; dental restoration; dental materials
MeSH Terms: conditions — Dental Plaque

INTERVENTIONS:
Procedure: dental restorative material surface preparation

SUMMARY:
In this study we intend to find out the pattern of biofilm accumulation in vivo on various surface finishings.

Our intention is to prepare Polymethylmetacrylate squers on orthodontical brackets,then prepare the surface of the sample and measure the surface roughness with a profilimeter and get the mean value in Ra units, then place the brackets on lower premolars and molars for 12 hours, remove them and examine the biofilm formed with confocal scanning microscope.

DETAILED DESCRIPTION:
Several studies in the past to assess the effects of surface roughness on the amount of plaque accumulation in vitro, whereas only few performed a modern in vitro assessment of the plaque accumulation. In this study we intend to find out the pattern of biofilm accumulation in vivo on various surface finishings.

Our intention is to prepare Polymethylmetacrylate squers on orthodontical brackets,then prepare the surface of the sample and measure the surface roughness with a profilimeter and get the mean value in Ra units, then place the brackets on lower premolars and molars for 12 hours, remove them and examine the biofilm formed with confocal scanning microscope.

Statistical evaluation of pilot study determined the need to perform this research on twelve(12) candidates. It is our intention to check two materials in each candidate: composite resin and polymethylmetacrylate.

ELIGIBILITY:
Inclusion Criteria:

* any patient with intact buccal surfaces of lower molars and premolars

Exclusion Criteria:

* patients that used antibiotics in the three months prior to the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-01; Study Completion 2006-08

PRIMARY OUTCOMES:
confocal scanning laser microscope evaluation of biofilm formation

SECONDARY OUTCOMES:
roughness analysis of the samples with profilometer

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Perez Davidi, DMD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Kawai K, Urano M, Ebisu S. Effect of surface roughness of porcelain on adhesion of bacteria and their synthesizing glucans. J Prosthet Dent. 2000 Jun;83(6):664-7. PMID 10842136
- See also: Michael Perez Davidi — http://www.mypd.co.il